CLINICAL TRIAL: NCT05780957
Title: Multi-Cancer Early Detection (MCED) of Firefighters
Status: Recruiting | Type: Observational
Sponsor: Vincere Cancer Center (Other)
Collaborators: Elypta (Industry); Proteotype (Unknown)
Responsible Party: Sponsor
Other Study IDs: VCC-MCEDFF-001
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Cancer; Multi-Cancer Early Detection; MCED
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighters who receive multi-cancer early detection (MCED) test
  Interventions: Other: MCED

INTERVENTIONS:
Other: MCED — multi-cancer early detection (MCED) test

SUMMARY:
This study is an an observational prospective cohort research study to explore the performance of new blood and urine tests for the early detection of cancer among firefighters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently employed as a firefighter, full-time or part-time
* Taking part in Vincere's First Responder Cancer Screening Program
* Able to donate blood and urine sample
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* Deemed medically unfit for sample donation
* Personal history of cancer in the last 5 years (with the exception of non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Actively working firefighters of any adult age, any gender and any demographic group are eligible, as well as no limitations regarding general health status other than those specified in the protocol Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive performance values (PPV and NPV) to detect cancer using Elypta's MCED test, as measured in plasma, in urine, and in plasma and urine combined | Up to 7 years
Sensitivity, specificity, positive and negative predictive performance values to detect cancer using Proteotype's MCED test, as measured in plasma. | Up to 2030

CONTACTS AND LOCATIONS:
Overall Officials: Vershalee Shukla, MD, Principal Investigator — Vincere Cancer Center
Locations (1):
- Vincere Cancer Center, Scottsdale, Arizona, United States